CLINICAL TRIAL: NCT06833008
Title: An Open-label, Phase I/II First-in-human, Dose Escalation and Confirmation Study to Evaluate the Safety, Tolerability, Pharmacokinetic, Pharmacodynamic and Anti-tumour Activity of IPN01195 as Single Agent in Adult Participants With Advanced Solid Tumours
Brief Title: A Study to Assess a New Medicine Called IPN01195 When Administered Alone in Adults With Advanced Solid Tumours
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-01195-450
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (dose escalation) (Experimental): IPN01195 will be administered at assigned dose level.
  Interventions: Drug: IPN01195
- Part B - (randomisation) (Experimental): Participants will be randomised to one of the two doses of interest once the PADR is determined
  Interventions: Drug: IPN01195

INTERVENTIONS:
Drug: IPN01195 — IPN01195 will be administered at assigned dose level.

SUMMARY:
The purpose of this study is to determine the appropriate dosage, safety and effectiveness of a new study drug IPN01195 in adults with advanced solid tumours.

The participants in this study will have advanced solid tumours. 'Advanced solid tumours' refers to cancers that can occur in several places, including cancers in organs or tissues that have spread from their original site to nearby tissues or other parts of the body.

DETAILED DESCRIPTION:
The study consists of two phases, called phase I and phase II.

Phase I will be conducted in two parts:

Part A: Phase I Part A study (dose escalation) is designed to find the dose range showing activity on the tumour that can be tolerated by the participants by testing different doses of IPN01195.

Part B: Phase I Part B of the study (dose confirmation) will assess the ability of study drug to prevent, slow down, or stop the growth of tumours (abnormal cell growths that can lead to cancer) and how the body processes and responds to the study drug when administered in a "low dose" or "high dose" and further explore the safety and tolerability.

These parts will consist of the following periods:

* A period to assess eligibility (screening period).
* A treatment period that will require at least two visits for the first month followed by one visit every month. There will be also one visit, at the end of treatment, at 30 days after the last administration of study drug.

An assessment visit will be required every 6 weeks up to Week 24 and every 12 weeks thereafter to measure the tumour again and to assess how it is evolving, whether it is getting bigger, smaller, is stable or has gone away.

Based on the results obtained from phase I, a phase II extension study will be included through to an updated study plan, to further evaluate the study drug.

In both study phases, participants will undergo blood samplings, urine collections, physical examinations and clinical evaluations. They may continue some other medications, but the details need to be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥18 years of age or the country's legal age of majority if the legal age is more than 18 years at the time of signing the informed consent.
* Participants with histologically confirmed metastatic solid tumour for whom no suitable alternative standard therapy exists.
* Participants must bear tumours harbouring selected classes of genetic alterations of MAPK pathway based on an analytically validated assay performed by an accredited laboratory.
* Part A: Participants must consent to the use of archival tumour tissue or, if not available, collection of fresh tumour biopsy at screening, for central confirmation of mutation status.
* Part B: Participants must consent to the use of archival tumour tissue or, if not available, collection of fresh tumour biopsy at screening, for MAPK genomic testing to confirm eligibility.
* Participants must have measurable disease per Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1
* Eastern Cooperative Oncology Group (ECOG)/performance status (PS) of 0 or 1
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Gastrointestinal conditions that could impair absorption of IPN01195 (specific cases e.g. remote history of gastrointestinal surgery, may be enrolled after discussion with the medical monitor)
* Any evidence of severe active infection or inflammatory condition.
* Non-adequate cardiac function
* Known psychiatric or substance abuse disorder, or any other cognitive disorder per the opinion of the investigator that would interfere with the participant's ability to cooperate with the requirements of the study.
* Underlying medical conditions that, in the investigator's or sponsor's opinion, will obscure the interpretation of toxicity determination or AEs.
* Known second malignancy either progressing or requiring active treatment within the last 2 years prior to first dose of the study intervention.
* Active brain metastases or leptomeningeal
* Current enrolment or past participation in any other clinical studies involving an investigational study treatment within the last 28 days
* Live vaccine(s) within 28 days prior to first dose of the study intervention or plan to receive such vaccines during the study.
* Concurrent treatment with any other anti-cancer therapy (including radiotherapy or investigational agents).
* Washout period of less than 28 days prior anti-cancer therapy (including chemotherapy, targeted agents, radiotherapy). If the participant was treated with an agent having a short half-life, washout can be <28 days but not shorter than 5 times the half-life.
* Condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 2 weeks prior to first dose of the study intervention.
* Non-adequate bone marrow function
* Non-adequate renal function
* Non-adequate hepatic function
* Known human immunodeficiency virus (HIV) infection. HIV testing will be performed in any countries where mandatory per local requirements.
* Known uncontrolled or untreated hepatitis infection.

  * (a) Known uncontrolled hepatitis B virus (HBV) infection.
  * (b) Known untreated current hepatitis C virus (HCV) infection.
* Sensitivity to IPN01195 or any of its components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2028-10-03 (Estimated); Study Completion 2028-10-03 (Estimated)

PRIMARY OUTCOMES:
Part A: Percentage of participants with dose limiting toxicity (DLT) | Part A: within 28 days of first dose.
Part A and B: Percentage of participants experiencing treatment emergent adverse events (TEAEs) and treatment emergent serious adverse events (TE SAEs). | From the first IPN01195 administration to 30 days after last dose.
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAE is an AE for which the start date is on or after the date that the intervention began.
Part A and B: Percentage of participants with dose interruptions and permanent treatment discontinuations | From the first study drug administration to 30 days after last dose.
Part B: Objective response rate (ORR) | Part B: At end of study (up to approximately 3 years)
  Objective response rate is defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) as determined by investigator per RECIST version 1.1.

SECONDARY OUTCOMES:
Part A: Time to maximum observed drug concentration (Tmax) after single and multiple doses of IPN01195 | Cycle 1: at Day 1 and at Day 15.
Part A: Maximum observed drug concentration (Cmax) after single and multiple doses of IPN01195 | Cycle 1: at Day 1 and at Day 15.
Part A: Area under the plasma concentration time curve (AUCtau) after single and multiple doses of IPN01195 | Cycle 1: at Day 1 and at Day 15.
  AUCtau is defined as the concentration of drug over one dosing interval.
Part A: Geometric mean ratio of Cmax of IPN01195 administered in fed state relative to fasted state. | Between Day -8 and Day -3 (fasted period) and between Day -10 and Day -7 (fed state period)
Part A: Geometric mean ratio of AUClast of IPN01195 administered in fed state relative to fasted state | Between Day -8 and Day -3 (fasted period) and between Day -10 and Day -7 (fed state period)
  AUClast is defined as the concentration of drug from time zero to the last observable concentration.
Part A: Geometric mean ratio of AUCinf of IPN01195 administered in fed state relative to fasted state | Between Day -8 and Day -3 (fasted period) and between Day -10 and Day -7 (fed state period)
  AUCinf is defined as the concentration of drug extrapolated to infinite time.
Part A: Prolongation of corrected QT interval (QTc) | Within 28 days of first dose.
  Prolongation of QTc defined as the upper limit of 90% confidence interval for change from baseline QTc evaluated over Cycle 1 at the highest clinically relevant exposure.
Part A: Objective response rate (ORR) | Part A: From first study drug administration to end of study (up to approximately 3 years)
  The ORR is defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) as determined by investigator per RECIST version 1.1
Part B: Duration of response (DoR) | Every 3 months until end of study or death (up to approximately 3 years)
  DoR defined as the time from first documented evidence of CR or PR until progressive disease, as determined by investigator per RECIST version 1.1.
Part B: Progression-free survival (PFS) | From first study drug administration to end of study (up to approximately 3 years)
  PFS is defined as the time from the date of first IPN01195 administration to the date of the first documented disease progression, as determined by investigator per RECIST version 1.1.
Part B: PFS rate at 4 months | At Month 4
  PFS rate at 4 months defined as the proportion of participants who remain alive and progression-free at 4 months, as determined by investigator per RECIST version 1.1.
Part B: Disease control rate (DCR). | Part B:From first study drug administration to end of study (up to approximately 3 years)
  DCR is defined as the percentage of participants with BOR of CR, PR or stable disease (SD), as determined by investigator per RECIST version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (13):
- United States (5):
  - START Mid-West, Grand Rapids, Michigan
  - Sarah Cannon Research Institute (SCRI) - Nashville, Nashville, Tennessee
  - Mary Crowley Cancer Research Centers - Medical City Hospital - Dallas, Dallas, Texas
  - START Mountan Region, West Valley City, Utah
  - Virginia Cancer Specialist- Fairfax, Fairfax, Virginia
- France (3):
  - Centre Léon Bérard - Lyon, Lyon
  - Paris Saint-Louis, Paris
  - IGR-Villejuif, Villejuif
- Italy (2):
  - Istituto Nazionale dei Tumori, Milan
  - Istituto Nazionale Tumori IRCCS - Fondazione Pascale, Napoli
- Spain (3):
  - Val D'Hebron, Barcelona
  - Hospital Universitario Quirónsalud Madrid, Madrid
  - M.D. Anderson Center Madrid, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/